CLINICAL TRIAL: NCT04398771
Title: A Multicenter, Single-arm, Prospective, Observational Study to Evaluate the Safety and Effectiveness of a Fixed-dose Combination Containing Valsartan and Rosuvastatin (Rovatitan® Tablet) in Patient With Hypertension and Hypercholesterolemia
Brief Title: To Evaluate Safety and Effectiveness of RovatitanTab.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: LG Chem (Industry)
Responsible Party: Sponsor
Other Study IDs: LG-VROS001
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Hypertension; Hyperlipidemias
MeSH Terms: conditions — Hypertension; Hyperlipidemias | interventions — Rosuvastatin Calcium; Valsartan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Rovatitan 5/80mg (Rosuvastatin 5mg/Valsartan 80mg) Rovatitan 5/160mg (Rosuvastatin 5mg/Valsartan 160mg) Rovatitan 10/80mg (Rosuvastatin 10mg/Valsartan 80mg) Rovatitan 10/160mg (Rosuvastatin 10mg/Valsartan 160mg) Rovatitan 20/80mg (Rosuvastatin 20mg/Valsartan 80mg) Rovatitan 20/160mg (Rosuvastatin 20mg/Valsartan 160mg)
  Interventions: Drug: Rosuvastatin/Valsartan

INTERVENTIONS:
Drug: Rosuvastatin/Valsartan — Rovatitan QD for 12 weeks
  Other Names: Rovatitan Tab.

SUMMARY:
To evaluate the safety and effectiveness of a fixed-dose combination containing valsartan and rosuvastatin (Rovatitan® Tablet) in patient with hypertension and hypercholesterolemia

DETAILED DESCRIPTION:
* Effectiveness: the ratio of patients who reach target BP or LDL-cholesterol
* Safety: we will collect safety data

ELIGIBILITY:
Inclusion Criteria:

* Patients who have hypertension and hyperlipidemia and older than 19 years
* Patients who undertstand purpose and method of study, agree with study

Exclusion Criteria:

* Patients who have been administered Rosuvastatin/Valsartan as a anti- hyperlipiddemic/anti-hypertensive drugs
* Uncontrolled hypertension (SBP>=180mmHg or DBP>=110mmHg)
* Patients who participated another clinical study or observational study 3 months ago.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have hypertension and hyperlipidemia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
The ratio of patients who reach the target BP | 12weeks
  SBP/DBP<140/90mmHg (<60years), SBP/DBP<150/90mmHg (>=60years)
The ratio of patients who reach the target LDLcholesterol | 12weeks
  target LDL refered to Hyperlipidemia pharmacotherapy

SECONDARY OUTCOMES:
The ratio of patients who reach the target BP and LDL-c | 12weeks
  SBP/DBP<140/90mmHg (<60years), SBP/DBP<150/90mmHg (>=60years), target LDL

CONTACTS AND LOCATIONS:
Overall Officials: Kang seokmin, Principal Investigator — Severance Hospital

IPD SHARING:
Plan to Share IPD: Undecided